CLINICAL TRIAL: NCT06544512
Title: Investigation of the Effect of Progressive Relaxation Exercises on Anxiety and Pain Level in Patients Undergoing Obesity Surgery
Brief Title: Effect of PMR on Anxiety and Pain Level in Patients Undergoing Obesity Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Şuheda Zorer, research assistant, Ataturk University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AtaturkUNI00
Record Dates: First submitted 2024-05-02; First posted 2024-08-09 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Anxiety; Pain, Postoperative
MeSH Terms: conditions — Anxiety Disorders; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: intervention and control
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the group that performed relaxation exercises (Experimental): The group that received progressive relaxation exercise and filled out the pain and state-trait anxiety scales
  Interventions: Other: progressive relaxation exercise
- the group that did not do relaxation exercises (No Intervention): The group that did not receive progressive relaxation exercise and only filled out the pain and state-trait anxiety scales

INTERVENTIONS:
Other: progressive relaxation exercise — looking at pain and anxiety by practicing progressive relaxation exercises
  Arms: the group that performed relaxation exercises

SUMMARY:
The aim of this clinical trial is to find out whether progressive relaxation exercises work on the effect of anxiety and pain level in patients undergoing obesity surgery. The main questions that it aims to answer are:

* Do progressive relaxation exercises reduce participants' pain levels?
* Do progressive relaxation exercises reduce participants' anxiety levels? The researchers will compare the effect of progressive relaxation exercises on the level of anxiety and pain between experimental and control groups .

Participants:

* He will experience obesity surgery surgery as planned for the first time

  * Who volunteered to participate in the research
* 18 years and over
* The mental state is healthy

DETAILED DESCRIPTION:
Obesity, which has been increasing in frequency in recent years, is a public health problem that many factors such as age, gender, education level, marital status and lack of physical activity are responsible for. The treatment of obesity can be divided into several stages: diet, physical activity, medical treatment and surgical treatment. Obesity surgery is resorted to in cases where diet therapy or medical treatment accompanied by physical activity does not give results. The sick individual is concerned both as a result of the physical effects of the disease on himself or as a result of the environmental change brought about by hospitalization. Encountering procedures that cause physical pain, being away from family, losing one's job, encountering unknown tools and procedures are some of the factors that may cause the hospitalized individual to feel anxiety. Having surgery is also among these factors and occupies an important place. Surgery includes the meanings of pain for the patient, loss of independence, deterioration in body image, and each of these elements is perceived as a threat. Nonpharmacological treatment to reduce postoperative pain and anxiety; the patient can be relieved by using methods such as diverting attention, listening to music, relaxation, breathing techniques, meditation, hypnosis. Progressive relaxation exercises are one of these methods. Progressive relaxation exercises involve the voluntary stretching and Novation of all muscle groups in the human body. Progressive relaxation exercise is a type of exercise that relaxes a person physically and spiritually, reduces a person's blood pressure, pain sensitivity, fatigue, stress, anxiety, heart rate, and positively affects a person physically and spiritually.The aim of this clinical trial is to find out whether progressive relaxation exercises work on the effect of anxiety and pain level in patients undergoing obesity surgery. The main questions that it aims to answer are:

* Do progressive relaxation exercises reduce participants' pain levels?
* Do progressive relaxation exercises reduce participants' anxiety levels? This research is planned to be conducted at the General Surgery Clinic of Van Yüzüncü Yıl University Dursun Odabaş Medical Center between August 2023- March 2024. The research is planned to be conducted in the General Surgery Clinic of Van Yüzüncü Yil University. Dependent Variables: State-Trait Anxiety scale, VAS Pain Scale Independent Variables: Training in progressive relaxation exercises Control Variables: the patient's age, gender, marital status, educational level, the status of having had surgery before, the status of having another health problem.

Collection of Data and Initiatives:Firstly, approval from the Ethics Committee of Atatürk University Faculty of Medicine and written permissions from the hospitals where the research will be conducted were obtained for the research. The "Patient Introduction Form", the "Condition-Continuity Anxiety Scale", the "Visual Analog Scale (VAS) Pain Form" will be used in the collection of research data. The data collection tools will be applied as follows: Questionnaires will be filled out by the researcher to the patients using the face-to-face interview technique.The scales will be introduced and the Patient Introduction form, the Status-Trait Anxiety Scale and the Visual Analog Scale (VAS) Pain Form will be completed. Later relaxation exercises will be performed during a session lasting 30 minutes, and after the session, the State-Trait Anxiety Scale and the Visual Analog Scale (VAS) Pain Form will be re-applied to patients.

ELIGIBILITY:
Inclusion Criteria:

* He will experience obesity surgery surgery as planned for the first time
* Who volunteered to participate in the research 18 years and over
* The mental state is healthy
* Without vision, hearing and speech problems
* Patients who know Turkish will be included in the study.

Exclusion Criteria:

* The patient has had bariatric surgery before,
* Have previously applied progressive relaxation exercises,
* Having a communication problem,
* Progressive relaxation exercise prevents the practice of health problems (epilepsy, bipolar disorder, schizophrenia, fever, infection, etc.) to be
* It has been determined that the patient does not want to be involved in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
VAS( Visual Analog Scale) | on the day of the surgery
  It is a scale with two different names on the two ends on a 10 cm long vertical or horizontal line (0=no pain, 10=most severe pain). The patient is asked to mark the point on this line that corresponds to the intensity of pain he feels.
State-Trait Anxiety Scale | on the day of the surgery
  The State-Trait Anxiety Inventory, which was adapted to Turkish culture by Öner and Le Compte (1983), and in which validity and reliability studies were conducted as well as norm studies, consists of a total of 40 items, including a State Anxiety Scale consisting of 20 items and a Trait Anxiety Scale consisting of 20 items. According to the "Item Remainder" correlation technique, which provides detailed information about the reliability and validity of the items forming the scale; the item reliability correlations of the Turkish form are between 0.34 and 0.72 for the Trait Anxiety Scale and between 0.42 and 0.85 for the State Anxiety Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yüzüncü Yıl University Dursun Odabaş Medical Center, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided